CLINICAL TRIAL: NCT01840761
Title: Delayed Vasospasm After Aneurysm With the Standardization Treatment of Traditional Chinese Medicine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010B030700029; 2010B030700029 (Other Grant/Funding Number: China Guangdong Provincial Science and Technology Agency)
Record Dates: First submitted 2011-12-12; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Aneurysm
Keywords: delayed vasospasm,; medicine,; standardization
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- herbal drug (Experimental): Traditional Chinese herbal drug
  Interventions: Drug: herbal drug
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: herbal drug
  Arms: herbal drug
Drug: placebo
  Arms: Placebo

SUMMARY:
Delayed vasospasm (DCVS) is the most serious complication of aneurysmal subarachnoid hemorrhage (aSAH) perioperative period ,the incidence rate up to 30% to 90%, and often can cause severe brain ischemia or brain damage of delayed ischemic and even lead to cerebral infarction, to be the main factor of deadly and severe disability . (aSAH) perioperative delayed vasospasm (CVS) is the bottleneck to restrict the long-term effect. Since there is no standard clinical treatment programs, limiting the advantages and characteristics of traditional Chinese medicine to play.Guangdong Provincial Hospital of TCM is the province's Medical Center encephalopathy, treated 100 brain aneurysm patients each year, more than 80 times craniotomies and surgical interventions , with a rich source of patiengs to carry out the study. In this study, on the basis studies on hemorrhagic stroke of a yin and yang syndrome and comprehensive treatment programe of the State 1995,the 15th research , in accordance with characteristics of the pathophysiology and understanding of cause and pathogenesis in aSAH perioperative period , through expert advice and review of the literature, under the guidance of Liu Maocai who isChinese medicine practitioners of Guangdong province , from diagnosis, diagnosis and treatment,prescription drugs, and other aspects of efficacy evaluation, developmenting a standardized treatment program of delayed CVS after aSAH . To evaluate the efficacy of the standardized program by prospective, randomized,controlled clinical trial,improving the postoperative results, reducting significantly the mortality and morbidity patients with cerebral aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 14-80 years old patients;
* Comply with the diagnostic criteria for Chinese and Western medicine;
* Comply with embolization of intracranial aneurysms or cranial aneurysm surgery indications;
* Preoperative Hunt and Hess grade of Ⅰ ~ Ⅳ; The first disease or previous history of stroke but no sequelae;
* Acceptance within 72h onset cranial aneurysm embolization or craniotomy aneurysm surgeon;
* Informed consent;

Exclusion Criteria:

* The age of 14 years of age or in patients over 80 years of age;
* By hypertension, a variety of blood diseases, amyloid angiopathy, cerebral arteritis, cerebral abnormal vascular network (moyamoya disease), brain tumor brain metastases as a result of bleeding;
* Associated with cardiovascular, liver and kidney and hematopoietic system of primary disease, mental illness;
* 72h of onset did not receive cranial aneurysm embolization or craniotomy for aneurysm surgery were;

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of DCVS after aneurysmal postoperative | 3 months
  after 3-months chinese medicine treatment, through evaluating the incidence of delayed vasospasm after cerebral aneurysms , to assess the efficacy of Chinese medicine

SECONDARY OUTCOMES:
1 month, 3 month mortality | 14days,1 month,3 month
  after 3-months chinese medicine treatment, through evaluating 1 month, 3 month mortality after cerebral aneurysms , to assess the efficacy of Chinese medicine

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Science and Technology Agency, Guangzhou, Guangdong, China

REFERENCES:
- See also: Related Info — http://www.gdhtcm.com